CLINICAL TRIAL: NCT06720493
Title: Functional Hemodynamic Assessment in Shocked Patients in the Pediatric Intensive Care Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osman Gamal Hassan, Functional hemodynamic assessment in shocked patients in the Pediatric Intensive Care Unit, Assiut University
Other Study IDs: assessment of shocked patients
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Shock
Keywords: hemodynamics; shocked patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: echocardiographic assessment of shocked patients to fluid administration — hemodynamic assessment of pediatric shocked patients using different modalities like echocardiography and electrical cardiometry
  Other Names: electrical cardiometry assessment of shocked patients

SUMMARY:
is to assess Functional hemodynamic status in shocked patients in the Pediatric Intensive Care Unit

DETAILED DESCRIPTION:
Shock is a leading cause of morbidity and mortality in pediatric patients worldwide (1, 2). The prevalence of sepsis and septic shock has been reported to be around 1-26% of shock cases with mortality rates ranging from 5 to 35% in hospitalized children globally (3, 4).

Appropriate fluid resuscitation is crucial in the management of children with shock (5). The current American College of Critical Care Medicine (ACCM), Pediatric Advanced Life Support (PALS), and Surviving Sepsis Campaign Guidelines have focused on the implementation of early and goal-directed fluid therapy (6, 7). Many studies have shown that mortality in pediatric patients with septic shock has been significantly decreased with aggressive fluid administration (8, 9). However, overzealous fluid administration can also lead to fluid overload (FO) and has been associated with complications such as acute respiratory distress syndrome (ARDS), which results in poor outcomes including increased hospital length of stay and mechanical ventilator days (10-13). As a result, in the recent decades, a more restrictive approach for fluid resuscitation has emerged in adults and children vs. the usual aggressive fluid therapy (14-16).

Traditional use of subjective findings such as pulse volume, capillary refill time, and clinical signs of hydration status to predict fluid responsiveness (FR) has been proven to be unreliable (17, 18).

While there is a growing body of the literature on the use of non-invasive devices for objective hemodynamic monitoring, there is a paucity of the literature related to the assessment of FR using these measures in children with shock (19).

Noninvasive monitoring techniques for the assessment of various cardiovascular parameters are increasingly accepted as the current medical practice. Electrical cardiometry (EC) is one such method for the determination of stroke volume (SV), cardiac output (CO), and other hemodynamic parameters and is based on changes in electrical conductivity within the thorax (20).

ICON® based on Electrical Cardiometry™ (EC) technology (Osypka Medical GmbH, Berlin, Germany) is a noninvasive, continuous hemodynamic monitoring device. It determines the CO by measuring variations in the thoracic electrical bioimpedance with phases of a cardiac cycle. During diastole, the erythrocytes in the aorta assume a random orientation (more impedance), while during systole the pulsatile blood flow causes them to align parallel to both the blood flow and the electrical current (less impedance). The magnitude of the maximum rate of change of impedance with a change in the orientation of erythrocytes gives a peak aortic blood flow acceleration and stroke volume (21).

Cardiac index (CI), systemic vascular resistance index (SVRI), cardiac contractility, stroke volume variation (SVV) and thoracic fluid content (TFC) are derived using complex mathematical formulae and patented algorithms. The accuracy and the clinical utility of electrocardiometry have been validated against other measures of CO like direct Fick' s method, thermodilution, and transthoracic and transesophageal echocardiography in a wide spectrum of patient conditions and populations across all ages, including critically ill patients, intraoperative settings, cardiac catheterization, and congenital heart diseases (22-26).

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 month and 18 years admitted to PICU with shock state
* Critically ill child who needs continuous hemodynamic monitoring in PICU

Exclusion Criteria:

* Age below one month of age and above 18 years
* Postoperative patients

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: shocked patients of age above one month and below 18 years
Sampling Method: Non-Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Functional hemodynamic assessment in shocked patients in the Pediatric Intensive Care Unit | baseline
  is to assess the need for fluid boluses administration in patients with shock

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566
- [Result] Lee SJ, Ramar K, Park JG, Gajic O, Li G, Kashyap R. Increased fluid administration in the first three hours of sepsis resuscitation is associated with reduced mortality: a retrospective cohort study. Chest. 2014 Oct;146(4):908-915. doi: 10.1378/chest.13-2702. PMID 24853382
- [Result] Davis AL, Carcillo JA, Aneja RK, Deymann AJ, Lin JC, Nguyen TC, Okhuysen-Cawley RS, Relvas MS, Rozenfeld RA, Skippen PW, Stojadinovic BJ, Williams EA, Yeh TS, Balamuth F, Brierley J, de Caen AR, Cheifetz IM, Choong K, Conway E Jr, Cornell T, Doctor A, Dugas MA, Feldman JD, Fitzgerald JC, Flori HR, Fortenberry JD, Graciano AL, Greenwald BM, Hall MW, Han YY, Hernan LJ, Irazuzta JE, Iselin E, van der Jagt EW, Jeffries HE, Kache S, Katyal C, Kissoon N, Kon AA, Kutko MC, MacLaren G, Maul T, Mehta R, Odetola F, Parbuoni K, Paul R, Peters MJ, Ranjit S, Reuter-Rice KE, Schnitzler EJ, Scott HF, Torres A Jr, Weingarten-Arams J, Weiss SL, Zimmerman JJ, Zuckerberg AL. American College of Critical Care Medicine Clinical Practice Parameters for Hemodynamic Support of Pediatric and Neonatal Septic Shock. Crit Care Med. 2017 Jun;45(6):1061-1093. doi: 10.1097/CCM.0000000000002425. PMID 28509730
- [Result] Weiss SL, Fitzgerald JC, Pappachan J, Wheeler D, Jaramillo-Bustamante JC, Salloo A, Singhi SC, Erickson S, Roy JA, Bush JL, Nadkarni VM, Thomas NJ; Sepsis Prevalence, Outcomes, and Therapies (SPROUT) Study Investigators and Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Global epidemiology of pediatric severe sepsis: the sepsis prevalence, outcomes, and therapies study. Am J Respir Crit Care Med. 2015 May 15;191(10):1147-57. doi: 10.1164/rccm.201412-2323OC. PMID 25734408
- [Result] de Souza DC, Shieh HH, Barreira ER, Ventura AM, Bousso A, Troster EJ; LAPSES Group. Epidemiology of Sepsis in Children Admitted to PICUs in South America. Pediatr Crit Care Med. 2016 Aug;17(8):727-34. doi: 10.1097/PCC.0000000000000847. PMID 27362850
- [Result] Martin K, Weiss SL. Initial resuscitation and management of pediatric septic shock. Minerva Pediatr. 2015 Apr;67(2):141-58. Epub 2015 Jan 21. PMID 25604591
- [Result] Mendelson J. Emergency Department Management of Pediatric Shock. Emerg Med Clin North Am. 2018 May;36(2):427-440. doi: 10.1016/j.emc.2017.12.010. Epub 2018 Feb 10. PMID 29622332